CLINICAL TRIAL: NCT00849888
Title: Phase I Serum-Free Cultured Thymus Transplantation in DiGeorge Anomaly, IND9836
Brief Title: Serum-Free Thymus Transplantation in DiGeorge Anomaly
Acronym: SerumFree
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The sponsor decided to withdraw the study.
Sponsor: Sumitomo Pharma Switzerland GmbH (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00006109; 1R01FD003528-01 (FDA); 2R01AI047040-11A2 (NIH); 5K12HD043494-09 (NIH); R01AI047040 (NIH); R01AI054843 (NIH); R56 Bridge R01AI4704011A1 (Other Grant/Funding Number: [NIH American Recovery and Reinvestment Act (ARRA) of 2009])
Record Dates: First submitted 2009-02-22; First posted 2009-02-24 (Estimated); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: DiGeorge Anomaly
Keywords: Thymus Transplantation; DiGeorge Anomaly; Athymia; Low T cell numbers; Immunoreconstitution; Immunodeficiency
MeSH Terms: conditions — DiGeorge Syndrome; Thymic aplasia; Immunologic Deficiency Syndromes | interventions — Immunosuppression Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atypical Complete DiGeorge (Experimental): Thymus Transplantation with Immunosuppression
  Interventions: Biological: Serum Free Thymus Transplantation with Immunosuppression
- Typical Complete DiGeorge (Experimental): Thymus Transplantation without Immunosuppression
  Interventions: Other: Serum Free Thymus Transplantation without immunosuppression

INTERVENTIONS:
Biological: Serum Free Thymus Transplantation with Immunosuppression — Cyclosporine pre-transplant (trough 180-220ng/ml) until naive T cells develop. Subjects >4,000/cumm T cells, pre-transplant methylprednisolone or prednisolone 1-2mg/kg/day. All subjects pre-transplant days -5,-4,-3: 3 doses 2mg/kg rabbit anti-thymocyte globulin. Thymus tissue (unrelated donor), donor, & donor's mother screened for safety. Transplant under general anesthesia into quadriceps. First 2 subjects, FBS cultured thymus is transplanted in 1 leg & serum free (SF) in other. After first 2 subjects >10% naïve T cells, 3rd receives only SF thymus. After 3rd subject >10%naive T cells, 4th subject transplanted. Thymus dose 4-18 grams/m2 body surface area. Thymus biopsy 8-12 weeks post-transplant. Skin biopsy at time of transplant & thymus biopsy. Followed by immune evaluations.
  Other Names: IND 9836; Thymus Tissue Transplant
  Arms: Atypical Complete DiGeorge
Other: Serum Free Thymus Transplantation without immunosuppression — Thymus tissue (unrelated donor), donor, & donor's mother screened for safety. Transplant under general anesthesia into quadriceps. First 2 subjects: FBS cultured thymus transplanted in 1 leg & serum free cultured thymus in other leg. After first 2 subjects have thymopoiesis in serum-free biopsy, >10% naïve T cells, 3rd subject receives only serum free cultured thymus. After 3rd subject >10% naive T cells, 4th subject receives transplant of only serum free cultured thymus. Dose 4-18grams/m2 body surface area. At time of transplant, skin biopsy. Allograft biopsy & skin biopsy done 8 to 12 weeks post-transplant. (Graft biopsy not done if subject medically unstable.) Post-transplant, subjects followed by immune evaluations, using blood samples, for two years.
  Other Names: IND 9836; Thymus Tissue Transplant
  Arms: Typical Complete DiGeorge

SUMMARY:
The study purpose is to determine if thymus tissue cultured in a serum-free (SF) solution is a safe and effective treatment for atypical and typical complete DiGeorge anomaly. [Funding Source - FDA OOPD]

DETAILED DESCRIPTION:
Complete DiGeorge anomaly is a congenital disorder characterized by athymia. Without successful treatment, patients remain immunodeficient and usually die by age 2 years. In "typical" complete DiGeorge subjects who have no T cells, thymus transplantation without immunosuppression has resulted in diverse T cell development and good T cell function. In "atypical" complete DiGeorge subjects who have no thymus, a rash, and some T cells that presumably developed extrathymically, thymus transplantation with immunosuppression has resulted in diverse T cell development and good T cell function. Thus far, thymus transplantation studies have used thymus cultured in fetal bovine serum (FBS medium). This protocol's purpose is to determine whether transplanted thymus cultured in serum free medium can safely support thymopoiesis and T cell reconstitution as does FBS medium cultured thymus tissue in DiGeorge anomaly subjects. This protocol includes 2 arms: atypical DiGeorge subjects who will receive immunosuppression and thymus transplantation; and, typical complete DiGeorge subjects who will receive thymus transplantation without immunosuppression. Serum free medium use would reduce concerns of animal product exposure including potential exposure to bovine spongiform encephalopathy(BSE).

ELIGIBILITY:
Thymus Recipients Inclusion:

Complete DiGeorge anomaly diagnosis

Must have one of following:

* congenital heart disease
* hypocalcemia requiring replacement
* 22q11 or 10p13 hemizygous
* CHARGE

Atypical Arm:

* Must have, or have had, rash. If rash present, skin biopsy must show T cells. If rash resolved, must have >50/cumm T cells; & <50/cumm naive T cells or <5% total
* PHA response must be <40000 counts per minute(cpm) on immunosuppression; or, <75000cpm off immunosuppression. PHA test must be done 2x
* CD45RA+CD62L+ CD3+ T cells must be <50/mm3; or, <5% of total CD3. Test must be done 2x

Typical Arm:

* PHA response <20 fold or <5,000cpm
* Circulating CD3+CD45RA+CD62L+T cells <50/mm3 or <5% total T cells
* 2 tests of T cells & PHA response must show similar results

Biological Mother Inclusion:

-Must be recipient's biological mother

Thymus Recipient Exclusion:

* Heart surgery <4 weeks pre-transplant or within 3 months post-transplant
* Rejection by surgeon or anesthesiologist as surgical candidates
* Lack of sufficient muscle tissue to accept transplant
* Medical condition does not allow to undergo a biopsy
* HIV
* CMV(>500 copies/ml blood by PCR on 2 tests)
* Ventilator dependence
* GVHD
* Maternal T cells >20% of total T cells
* Prior immune reconstitution attempts (e.g., BMT, prior thymus transplant)
* Hypoparathyroidism meeting criteria for combined thymus/parathyroid transplant & parents desiring it
* RSV or parainfluenza virus
* Enterovirus or Adenovirus in stool

Biological Mother Exclusion:

-Unwillingness to sign consent or provide blood/buccal samples

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2008-04; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Survival | One year post-thymus transplantation.
  Survival at one year post thymus transplantation.
Incidence of graft-versus-host-disease (GVHD). | One year post-thymus-transplantation.
  Development of graft versus host disease in first year after transplantation associated with T cells from the thymus donor.
Thymopoiesis or graft rejection on biopsy. | Two months post-thymus transplantation.
  Graft rejection analysis by biopsy at 2 months post-thymus transplantation.

SECONDARY OUTCOMES:
Incidence of autoimmune disease. | By two years post-thymus transplantation.
  Incidence of autoimmune disease by year 2 after transplantation Cytopenias as assessed by complete blood counts and differential. Thyroid disease as assessed by thyroid function tests
Immune outcomes: T cell development; evaluate T cell numbers, diversity, and function. | One year post-thymus transplantation.
  Number of naïve CD4 T cells at one year after transplantation Number of total CD4 T cells at one year after transplantation Proliferative response to PHA at one year after transplantation TCRBV diversity by spectratyping measured by DKL score at one year after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: M. Louise Markert, M.D., Ph.D, Principal Investigator — Duke University Medical Center, Pediatrics, Allergy & Immunology

REFERENCES:
- [Background] Markert ML, Devlin BH, Alexieff MJ, Li J, McCarthy EA, Gupton SE, Chinn IK, Hale LP, Kepler TB, He M, Sarzotti M, Skinner MA, Rice HE, Hoehner JC. Review of 54 patients with complete DiGeorge anomaly enrolled in protocols for thymus transplantation: outcome of 44 consecutive transplants. Blood. 2007 May 15;109(10):4539-47. doi: 10.1182/blood-2006-10-048652. Epub 2007 Feb 6. PMID 17284531
- [Background] Markert ML, Alexieff MJ, Li J, Sarzotti M, Ozaki DA, Devlin BH, Sedlak DA, Sempowski GD, Hale LP, Rice HE, Mahaffey SM, Skinner MA. Postnatal thymus transplantation with immunosuppression as treatment for DiGeorge syndrome. Blood. 2004 Oct 15;104(8):2574-81. doi: 10.1182/blood-2003-08-2984. Epub 2004 Apr 20. PMID 15100156
- [Background] Markert ML, Sarzotti M, Ozaki DA, Sempowski GD, Rhein ME, Hale LP, Le Deist F, Alexieff MJ, Li J, Hauser ER, Haynes BF, Rice HE, Skinner MA, Mahaffey SM, Jaggers J, Stein LD, Mill MR. Thymus transplantation in complete DiGeorge syndrome: immunologic and safety evaluations in 12 patients. Blood. 2003 Aug 1;102(3):1121-30. doi: 10.1182/blood-2002-08-2545. Epub 2003 Apr 17. PMID 12702512
- [Background] Selim MA, Markert ML, Burchette JL, Herman CM, Turner JW. The cutaneous manifestations of atypical complete DiGeorge syndrome: a histopathologic and immunohistochemical study. J Cutan Pathol. 2008 Apr;35(4):380-5. doi: 10.1111/j.1600-0560.2007.00816.x. PMID 18333898
- [Background] Chinn IK, Devlin BH, Li YJ, Markert ML. Long-term tolerance to allogeneic thymus transplants in complete DiGeorge anomaly. Clin Immunol. 2008 Mar;126(3):277-81. doi: 10.1016/j.clim.2007.11.009. Epub 2007 Dec 26. PMID 18155964
- [Background] Markert ML, Li J, Devlin BH, Hoehner JC, Rice HE, Skinner MA, Li YJ, Hale LP. Use of allograft biopsies to assess thymopoiesis after thymus transplantation. J Immunol. 2008 May 1;180(9):6354-64. doi: 10.4049/jimmunol.180.9.6354. PMID 18424759